CLINICAL TRIAL: NCT07401563
Title: Enhancing Community Participation and Service Access for Transitional-Age Youth and Young Adults With Developmental Disabilities Through Community Mobility Plans
Brief Title: Community Mobility Plans: Improving Community Participation Through Travel Interventions for Adolescents and Young Adults With Intellectual and Developmental Disabilities
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31078; 901FDV0034-01-00 (Other Grant/Funding Number: Field Initiated Project, National Institute in Disability, Independent Living, and Rehabilitation Research (NIDILRR))
Record Dates: First submitted 2026-01-23; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Intellectual and Developmental Disability
Keywords: Community Mobility; Young Adults; Adolescents; Transportation; Community Mobility Planning; Travel Intervention
MeSH Terms: conditions — Developmental Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Community Mobility Planning Process (Experimental)
  Interventions: Behavioral: Community Mobility Planning Process (CMPP)

INTERVENTIONS:
Behavioral: Community Mobility Planning Process (CMPP) — The Community Mobility Planning Process (CMPP) consists of 5 steps to be implemented over an 8-week period. The steps take a young adult with intellectual or developmental disabilities and their support staff through a series of activities to help them develop a plan to be more independent in their daily activities. Step 1: Identify Person-Centered Community Mobility Priorities & Preferences (Weeks 1-4), Step 2: Evaluate Person & Environment Components Supporting Community Mobility (Weeks 5-8), Step 3: Set a Person-Centered Community Mobility Goal (Weeks 9-10), Step 4: Deliver Interventions to Support Community Mobility (Weeks 11-21), Step 5: Evaluate Progress (Weeks 22-24). Each step has objectives and activities to support learning.

SUMMARY:
The goal of this study is to establish a proof-of-product by evaluating and refining the "Community Mobility Planning Process" curriculum activities with adolescents and young adults (AYA; ages 16-25 years) with Intellectual Disabilities (ID).

The main questions it aims to answer are:

- Is the Community Mobility Planning Process feasible to implement with adolescents and young adults with ID?

Participants will:

* Complete surveys and patient-reported outcome measures (PROMs) related to their experiences, attitudes, and feelings about community mobility.
* Complete a series of structured activities including worksheets, discussions, and specific skill building activities and share de-identified worksheets with the research team.
* Provide feedback about what they liked and didn't like about the the Community Mobility Planning Process.

ELIGIBILITY:
Inclusion Criteria:

* Part of the program/classroom where professional plans to implement the Community Mobility Planning Process.
* 16-30 at start of implementation.
* Mild to moderate intellectual disability.
* Can participate in program activities in English.

Exclusion Criteria:

* Plan to end/stop participation in the current organization in <9 months from time of enrollment.
* A developmental disability without an intellectual disability
* Participants considered legally blind or deaf will be excluded to ensure a more homogeneous group for the initial development process

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Community Mobility Experience | Pre-test, 1 month Post-test
  This survey assesses how often and how easily individuals with intellectual and developmental disabilities (IDD) leave home to participate in daily activities. It includes questions on transportation use, satisfaction, ease of access, and barriers or supports to community mobility. Responses help inform transportation needs and evaluate mobility-related interventions. The Community Mobility Experience Survey includes four scoring domains: frequency of community mobility (1-5), ease of mobility (1-4), sufficiency of mobility (0-2), and satisfaction with mobility (1-4). Higher scores indicate greater frequency, ease, sufficiency, or satisfaction with community mobility. In addition, specific transportation modes are evaluated across the same four domains-frequency, ease, sufficiency, and satisfaction-using the same scoring scales.
Community Mobility Self-Efficacy | Pre-test, 1 month Post-test
  This brief self-report measure assesses an individual's confidence in completing key steps related to community mobility and transportation planning. The scale responses are informed by standards outline by Bandura's self-efficacy theory, and items are modified from the general self-efficacy scale. Scores range from 20 to 60, with higher scores indicating a greater feeling of self-efficacy with community mobility.
PROMIS Satisfaction with Participation and Discretionary Social Activities | Pre-test, 1 month Post-test
  This brief PROM, available from PROMIS, evaluates satisfaction with level of involvement in leisure activities. Scores range from 7 to 35, with higher scores indicating higher satisfaction with social roles and activities.

CONTACTS AND LOCATIONS:
Overall Officials: Beth Pfeiffer, PhD, OTR/L, BCP, FAOTA, Principal Investigator — Temple University; Jessica Kramer, PhD, OTR/L, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No